CLINICAL TRIAL: NCT02015559
Title: Phase II Randomized Trial of Mugard Compared With Best Supportive Care for Prevention and Treatment of Stomatitis in Women With Hormone Receptor Positive Breast Cancer Initiating Treatment With Everolimus-based Endocrine Therapy.
Brief Title: Mucoadhesive Oral Wound Rinse in Preventing and Treating Stomatitis in Patients With ER- or PR-Positive Metastatic or Locally Recurrent Breast Cancer That Cannot be Removed by Surgery Receiving Everolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-001676; NCI-2013-02384 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TRIO-US B10 (Other: JonssonCCC)
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2019-05

CONDITIONS: Estrogen Receptor-positive Breast Cancer; HER2-negative Breast Cancer; Oral Complications; Progesterone Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (mucoadhesive oral wound rinse) (Experimental): Patients receive mucoadhesive oral wound rinse PO as a gentle swish for 30-60 seconds 3-6 times daily beginning on day 1 of everolimus therapy and continuing for up to 6 months in the absence of unacceptable toxicity.
  Interventions: Drug: mucoadhesive oral wound rinse; Other: laboratory biomarker analysis
- Arm II (no intervention) (No Intervention): Patients receive no intervention.

INTERVENTIONS:
Drug: mucoadhesive oral wound rinse — Given PO
  Other Names: MuGard; oral mucoadhesive protectant rinse
  Arms: Arm I (mucoadhesive oral wound rinse)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I (mucoadhesive oral wound rinse)

SUMMARY:
This randomized phase II trial studies how well mucoadhesive oral wound rinse works in preventing and treating stomatitis in patients with estrogen receptor (ER)- or progesterone receptor (PR)-positive metastatic or locally recurrent breast cancer that cannot be removed by surgery receiving everolimus. Mucoadhesive oral wound rinse may help prevent symptoms of stomatitis, or mouth sores, in patients receiving everolimus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate whether use of prophylactic MuGard (mucoadhesive oral wound rinse) in participants being treated with everolimus will reduce the rate of stomatitis.

SECONDARY OBJECTIVES:

I. Compare symptoms from mouth sores in patients receiving MuGard compared with those receiving best supportive care.

II. Evaluate the rate of everolimus dose adjustment or therapy discontinuation as a result of stomatitis in participants treated with MuGard prophylaxis versus best supportive care.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive mucoadhesive oral wound rinse orally (PO) as a gentle swish for 30-60 seconds 3-6 times daily beginning on day 1 of everolimus therapy and continuing for up to 6 months in the absence of unacceptable toxicity.

ARM II: Patients receive no intervention.

After completion of study treatment, patients are followed up within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally recurrent unresectable breast cancer
* Histological or cytological confirmed ER and/or PR positivity
* Progression through at least one prior line of endocrine therapy
* Participant is scheduled to initiate treatment with everolimus combined with exemestane or another form of endocrine therapy
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hgb) ≥>= 8.0 g/dL
* International normalized ratio (INR) =< 2
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 X upper limit of normal (ULN) (or =< 5 X ULN if hepatic metastases are present)

Exclusion Criteria:

* Human epidermal growth factor receptor 2 (HER2)-overexpressing breast cancer by local laboratory testing (immunohistochemistry [IHC] 3+ staining or fluorescent in situ hybridization [FISH] positive)
* Baseline presence of oral ulcers
* Prior treatment with everolimus or another mammalian target of rapamycin (mTOR) inhibitor (temsirolimus)
* Patients on warfarin (patients on injectable blood thinners, such as Lovenox, are able to continue those)
* Patients currently receiving chemotherapy or who have received chemotherapy less than 4 weeks of the start of everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by hemoglobin A1c (HbA1c) > 8% despite adequate therapy; patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Patients who have any severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction =< 6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Symptomatic congestive heart failure of New York heart Association class III or IV
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B virus surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA])
  * Known severely impaired lung function (spirometry and diffusing capacity of the lung for carbon monoxide [DLCO] 50% or less of normal and oxygen [O2] saturation 88% or less at rest on room air)
  * Active, bleeding diathesis
* Chronic treatment with corticosteroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed
* Known history of human immunodeficiency virus (HIV) seropositivity
* Patients who have received live attenuated vaccines within 1 week of start of everolimus and during the study; patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after; highly effective contraception methods include combination of any two of the following:

  * Use of oral, injected or implanted hormonal methods of contraception or
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository
  * Total abstinence or
  * Male/female sterilization Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of grades 1-4 stomatitis assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 7 days after completion of treatment
  Will be estimated and the 95% confidence interval (CI) will also be obtained. Chi-square test will be used to compare the stomatitis rates between the two study arms.

SECONDARY OUTCOMES:
Rate of grade 3/4 stomatitis assessed using CTCAE version 4.03 | Up to 7 days after completion of treatment
  Will be estimated and the 95% CI will also be obtained. Chi-square test will be used to compare the stomatitis rates between the two study arms.

OTHER OUTCOMES:
Rate of everolimus dose adjustment or discontinuation related to stomatitis | Up to 7 days after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Parvin Peddi, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States